CLINICAL TRIAL: NCT00513942
Title: Effects of Fetal Movement Counting - a Randomized Controlled Trial of an Unselected Population
Brief Title: Effects of Fetal Movement Counting in Third Trimester of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Responsible Party: Principal Investigator, Frederik Froen, Head of Department, Norwegian Institute of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NIPH-EPAM-335
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Decreased Fetal Movements, Unspecified Trimester, Other Fetus; Worries; Pregnancy
Keywords: Fetal Movement; Maternal-Fetal-Attachment; Fetus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (No Intervention): These women will follow standard antenatal care according to the Norwegian Guidelines
- B (Active Comparator): Intervention group for Fetal Movement Counting
  Interventions: Other: Fetal Movement Counting

INTERVENTIONS:
Other: Fetal Movement Counting — Women in the intervention group will receive an information pamphlet. The main items will be basic information and interpretation of fetal activity and instructions when to contact health professionals if experiencing DFM.
  Arms: B

SUMMARY:
The aim is to test effects of using formal kick counting chart in the third trimester of pregnancy in an unselected population. The research questions are:

Does Fetal Movement Counting (FMC):

1. Improve the identification of risk pregnancies/pathology?
2. Affect the women's well-being?
3. Stimulate maternal-fetal attachment antepartum?

DETAILED DESCRIPTION:
Fetal activity serves as an indirect measure of central nervous system integrity and function, and regular FM can be regarded as an expression of fetal well-being.A hypoxic fetus responds automatically by redistributing blood away from the non-essential organs which lead to a reduction of non-vital activities; movements. Conversely, pregnancies in which the mother report decreased fetal movements (DFM) is associated with adverse outcomes and may indicate danger for the fetus. In cases were DFM are associated with complications of pregnancy, maternal lack of sensitivity and awareness to fetal movements may be a risk factor for her pregnancy. The most important current identifier of DFM is the women's perception of what is a decrease of FM. Fetal movement counting may be a tool for the mothers that might increase identification of risk pregnancies.

The outcome measures are (referring to the research questions above):

1. Identification of risk pregnancies/pathology?

   1. Primary outcome measures: Numbers of identified pathological conditions in pregnancies (fetal growth restriction (FGR), acute caesarean section on fetal indication/non-reactive non-stress test (NST), oligohydramnios, pathologic blood flow in arteria umbilicalis, maternal perception of absent fetal movements for more than 24 hours before admission to hospital, or perinatal death).
   2. Secondary outcome measures: Frequency of consultations because of maternal concern, use of resources in evaluation of these pregnancies (NST, ultrasound, Doppler, recurrent consultations), induced or spontaneous start of delivery, mode of birth.
2. Affect the women's well-being?

   1. Primary outcome measure: Maternal concern.
   2. Secondary outcome measure: Maternal satisfaction with use of FMC and sense of control in interpretation of signals from own body and child.
3. Stimulate maternal-fetal attachment antepartum?

   1. Primary outcome measure: Maternal-fetal attachment.
   2. Secondary outcome measure: Health promoting behavior in pregnancy (smoking habits, use of alcohol, attending standard program for antenatal care).

ELIGIBILITY:
Inclusion Criteria:

* women booking at screening ultrasound in pregnancy week 17-20
* native speaking women
* singleton pregnancies

Exclusion Criteria:

* women with pregnancies with severe anomalies or other cause to consider termination

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2007-08; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Identification of pathological conditions in pregnancies and birth, maternal concern (Cambridge Worry Scale), maternal-fetal attachment (Prenatal Attachment Inventory) | One and a half year

SECONDARY OUTCOMES:
Frequency of consultations, use of resources and mode of birth, maternal satisfaction and sense of control in interpretation of signals from own body and child, health promoting behavior | One and a half year

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Froen, MD, PhD, Principal Investigator — Norwegian Institute of Public Health; Eli Saastad, CNM, MSc, Study Chair — Oslo and Akershus University College
Locations (1):
- Norwegian Institute of Public Health, Oslo, Norway

REFERENCES:
- [Derived] Saastad E, Winje BA, Stray Pedersen B, Froen JF. Fetal movement counting improved identification of fetal growth restriction and perinatal outcomes--a multi-centre, randomized, controlled trial. PLoS One. 2011;6(12):e28482. doi: 10.1371/journal.pone.0028482. Epub 2011 Dec 21. PMID 22205952
- [Derived] Winje BA, Saastad E, Gunnes N, Tveit JV, Stray-Pedersen B, Flenady V, Froen JF. Analysis of 'count-to-ten' fetal movement charts: a prospective cohort study. BJOG. 2011 Sep;118(10):1229-38. doi: 10.1111/j.1471-0528.2011.02993.x. Epub 2011 May 18. PMID 21585644